CLINICAL TRIAL: NCT07128745
Title: Developing, Implementing and Evaluating of Self-management Behavior Intervention Through Shared Medical Appointment for COPD Patients (SMA-COPD): a Multi-stage Mixed Methods Research
Brief Title: Shared Medical Appointment for COPD Patients (SMA-COPD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025YLSD No. 220-01
Record Dates: First submitted 2025-07-23; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD
Keywords: COPD; co-design; mixed methods; cluster randomized controlled trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Shared Medical Appointments

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study. Due to the nature of the intervention, participants, care providers, and investigators will be aware of group assignments. However, outcome assessors and data analysts will be blinded to participant group allocation to minimize the risk of bias during data evaluation and interpretation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared medical appointment with self-management behavior intervention strategy (Experimental): Shared medical appointment with self-management behavior intervention strategy. In each intervention community center, the 14 enrolled patients will be divided into two subgroups and receive shared medical appointment interventions.
  Interventions: Behavioral: Shared Medical Appointment + Self-Management Strategy
- Usual care with self-management handbook (Active Comparator): General practitioners will provide usual care to patients based on the standard consultation duration and distribute a COPD health education and behavioral guidance manual.
  Interventions: Behavioral: Usual Care + Self-Management Handbook

INTERVENTIONS:
Behavioral: Shared Medical Appointment + Self-Management Strategy — Participants assigned to this arm will receive a self-management intervention delivered through shared medical appointments (SMAs). The SMA intervention will be conducted once every two months for a total of three sessions over six months. Each session includes structured medical consultation, health education, behavioral guidance based on the Behavior Change Wheel (BCW) framework, and facilitated peer discussion.
  Arms: Shared medical appointment with self-management behavior intervention strategy
Behavioral: Usual Care + Self-Management Handbook — Participants receive routine one-on-one GP care plus a printed COPD self-management education handbook.
  Arms: Usual care with self-management handbook

SUMMARY:
The goal of this clinical trial is to evaluate whether a behavior change intervention, delivered through a shared medical appointment (SMA) model, can improve self-management behaviors and health outcomes among community-based patients with chronic obstructive pulmonary disease (COPD). The main questions it aims to answer are:

i) Can a BCW-based intervention strategy that integrates shared medical appointments increase COPD patients' self-management behaviors? ii) Does this strategy relate to reduced acute exacerbations, slower lung function decline, and improved health-related quality of life?

Researchers will compare the shared medical appointment group and the usual care group to see if integrating SMA improves behavioral and clinical outcomes.

Participants will i) Take part in group-based shared medical appointments once every two months for a total of three sessions over six months, led by a general practitioner, involving structured medical consultation, behavioral guidance, and peer interaction.

ii) Receive behavioral intervention based on the Behavior Change Wheel (BCW) framework, targeting modifiable factors influencing self-management behaviors.

iii) Complete questionnaires and assessments at baseline and 6-month follow-up to evaluate changes in behavior, symptoms, and quality of life.

The study uses a three-stage mixed methods design:

i) Stage 1 involves longitudinal qualitative interviews and co-design with patients and clinicians to develop the intervention strategy.

ii) Stage 2 is a pilot study to test the feasibility and acceptable for up-coming cluster randomized controlled trial.

iii)Stage 3 is a cluster randomized controlled trial to evaluate the effectiveness and mechanisms of the intervention.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) affects nearly 100 million patients in China, with poor self-management behaviors contributing to frequent exacerbations and increased disease burden. Despite inclusion in national basic public health services, limited healthcare resources hinder effective COPD management. Shared medical appointments (SMAs) offer a promising solution by providing group-based clinical care and behavioral interventions. This study aims to develop and evaluate a behavioral intervention strategy incorporating SMAs for community-based COPD self-management.

This multi-stage mixed methods study comprises three phases. Stage 1 uses patient-provider co-design and longitudinal qualitative research methods to analyze self-management behavioral factors based on the Behavior Change Wheel theory and develop the SMA-COPD intervention. Stage 2 conducts a feasibility study to assess intervention acceptability and research procedures. Stage 3 implements a cluster randomized controlled trial across 20 community health centers, recruiting 280 COPD patients (14 per cluster, 140 per arm). The intervention group receives three monthly SMA sessions, while controls receive routine care. Primary outcomes include COPD self-management behaviors, inhaler medication adherence, and health-related quality of life. Secondary outcomes include inhaler technique, lung function, physical activity capacity, and number of acute exacerbations. Data collection occurs at baseline and 6 months post-intervention, with additional assessments at 6 months post-intervention completion. The study follows the RE-AIM framework to evaluate reach, effectiveness, adoption, implementation, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for Chronic Obstructive Pulmonary Disease (COPD) according to the GOLD 2024 guidelines.
* Diagnosed with COPD within the past year, or has had fewer than two outpatient visits for COPD management in the past year.
* Resides in the community under the jurisdiction of the respective community health service centre.
* Aged 40 to 80 years.
* Has full cognitive and behavioural capacity and is able to clearly express personal will.
* No plans for long-term travel in the next six months.
* Has provided written informed consent and voluntarily agreed to participate in the study.

Exclusion Criteria:

* Has severe complications or other serious diseases.
* Has limited physical activity due to comorbidities or complications.
* Is currently participating in another clinical trial.
* Is unsuitable for participation by the study investigators.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-management behaviour | 6 months after intervention
  COPD self-management Scale. This scale comprises five dimensions: symptoms, daily life, emotions, information, and self-efficacy, with a total of 51 items. Each item is scored using a 5-point Likert scale, where higher scores indicate better performance in the patient's self-management behaviors.
  Zhang, C. H., He, G. P., Li, J. P., et al. (2011). Development and evaluation of a self-management scale for patients with chronic obstructive pulmonary disease. Chinese General Practice, 2011, 14(28), 3219-3223.
medication adherence | 6 months after intervention
  Scale of Test of the Adherence to Inhalers (TAI). Meng, W. W., Cui, Y. N., Luo, L. J., et al. (2022). The TAI questionnaire consists of 10 items, all of which are scored using a 5-point Likert scale, where 1 point indicates "always" and 5 points indicates "never." The total score ranges from 10 to 50, with lower scores indicating poorer adherence to inhaled medication in patients. Reliability and validity of the Chinese version of the Inhaler Adherence Test. Chinese Journal of Tuberculosis and Respiratory Diseases, (05), 423-430.
Quality of life of patients using SGRQ | 6 months after intervention
  The St George's Respiratory Questionnaire (SGRQ) is used to assess the severity of illness in patients with pulmonary diseases. It consists of 76 items (50 items in the U.S. version) divided into three domains: Symptoms, Activity, and Impacts on Daily Life. The scoring method employs a weighted average, where higher weights indicate a more severe impact on quality of life. The minimal clinically important difference (MCID) for this questionnaire is 4 points.

SECONDARY OUTCOMES:
Correct use of inhaled medication devices | 6 months after intervention
  Assessed using a 10-step inhaler technique evaluation checklist adapted from Qin Qiong et al. (2016), with each step scored as 1 point for a total of 10 points, where higher scores indicate better performance in using of inhaled medication devices.
Forced expiratory volume in one second, FEV1. | 6 months after intervention
  FEV1 (Forced Expiratory Volume in the first second) is the maximum volume of air exhaled in the first second after a maximal inhalation, measured during a forced expiratory maneuver. It is one of the most critical indicators in pulmonary function testing. FEV1 is commonly used to assess the severity of lung function impairment in conditions such as bronchial asthma and chronic obstructive pulmonary disease (COPD). Additionally, it can be combined with FVC (Forced Vital Capacity, the maximum volume of air exhaled forcefully after a full inhalation) to diagnose COPD. For instance, a post-bronchodilator FEV1/FVC ratio < 70% of the predicted value confirms a diagnosis of COPD.
Six-minute walk test distance | 6 months after intervention
  The 6-minute walk distance (6MWD) will be measured according to the American Thoracic Society (ATS) guidelines to evaluate functional exercise capacity in people with COPD. Greater walking distance indicates better cardiopulmonary function in patients.
Frequency of acute exacerbations requiring hospitalisation | 6 months after intervention
  Number of acute exacerbations requiring hospital readmission
Knowledge of COPD | 6 months after intervention
  COPD knowledge will be evaluated using the Bristol COPD Knowledge Questionnaire (BCKQ). The BCKQ assesses knowledge across 13 key domains: COPD etiology, epidemiology, symptoms, vaccination, smoking, infections, oral/inhaled corticosteroid therapy, exercise, antibiotics, and inhaled bronchodilators. Each domain contains 5 items (65 total items), with three response options per item: "True," "False," and "Don't know." Correct answers score 1 point; higher total scores indicate better COPD-related knowledge.
Beliefs About Medicines | 6 months after intervention
  The beliefs about medication will be assessed using the Beliefs about Medicines Questionnaire-Specific (BMQ-Specific). The BMQ-Specific assesses medication concern beliefs and necessity beliefs, each measured by 5 items with scores ranging from 5 to 25. Higher scores indicate stronger beliefs in the respective dimension.
Self-Efficacy | 6 months after intervention
  Self-efficacy will be assessed using the COPD Self-Efficacy Scale (CSES). The CSES comprises five dimensions: dyspnea management, emotional distress, physical activity, environmental/temperature factors, and safety behaviors, with a total of 31 items. Each item is rated on a 5-point Likert scale (1-5), where 1 = "not confident at all" and 5 = "very confident." Higher total scores indicate greater self-efficacy in patients during physical activities.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Haidian District Huayuan Road Community Health Service Centre, Beijing

IPD SHARING:
Plan to Share IPD: Yes
The data that support the publication will be shared with the publication.
Supporting Information: CSR
Time Frame: When the data analysis completed and the related paper published, the IPD and supporting information will be available for 3 years.
Access Criteria: IPD and supporting documents (e.g., study protocol, statistical analysis plan) will be available to qualified researchers upon reasonable request, subject to approval by the study steering committee.
  Accessible Data: De-identified IPD, including demographics, clinical outcomes, and behavioral intervention records, will be shared.
  Access Process: Requests should be submitted via email to the corresponding author, with a detailed research proposal and ethical approval proof. Data will be transferred through secure platforms after signing a data use agreement.